CLINICAL TRIAL: NCT06799533
Title: AN OPEN-LABEL PHASE 1 STUDY TO INVESTIGATE PF-08046031 IN ADULTS WITH ADVANCED MELANOMA AND OTHER SOLID TUMORS
Brief Title: A Study to Learn About the Study Medicine Called PF-08046031 in Advanced Melanoma and Other Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C5901001; 2024-514745-10-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Malignant Melanoma; Melanoma; Metastatic Melanoma; Solid Tumors
Keywords: Solid tumors; Other Solid tumors
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: single group assignment
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PF-08046031 monotherapy (Experimental): PF-08046031
  Interventions: Drug: PF-08046031

INTERVENTIONS:
Drug: PF-08046031 — Given into the vein (IV; intravenous)

SUMMARY:
This study will test the safety of a drug called PF-08046031 in participants with melanoma and other solid tumors that have no current approved treatment or have spread through the body. It will also study the side effects of this drug. A side effect is anything a drug does to the body besides treating the disease. The study will have 3 parts. Part A and B of the study will find out how much PF-08046031 should be given to participants. Part C will use the information from Parts A and B to see if PF-08046031 is safe and if it works to treat solid tumor cancers.

ELIGIBILITY:
Inclusion Criteria:

* Participants in Part 1 (dose escalation) must have histologically- or cytologically-confirmed metastatic or unresectable cutaneous melanoma. They must have progressive disease following at least 1 prior anti programmed death-1 (PD 1)/programmed death-ligand 1 (PD L1) immunotherapy containing regimen (either as monotherapy, or in combination with other checkpoint inhibitors or other therapies) and should have no appropriate standard therapy available at the time of enrollment in the judgment of the investigator.
* Participants in Part 2 (dose optimization) must have histologically- or cytologically-confirmed metastatic or unresectable cutaneous melanoma. They must have progressive disease following at least 1 prior anti PD 1/PD L1 immunotherapy containing regimen (either as monotherapy, or in combination with other checkpoint inhibitors or other therapies) but not more than 2 total prior lines of systemic therapy and should have no appropriate standard therapy available at the time of enrollment in the judgment of the investigator.
* For Part 3 (dose expansion): Participants must have histologically- or cytologically confirmed metastatic or unresectable solid malignancy from 1 of the following tumor types: cutaneous melanoma, NSCLC, HNSCC, esophageal cancer.

Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1 Measurable disease per RECIST v1.1 at baseline

• Participants who have refused available standard of care therapies are not eligible.

Exclusion Criteria:

• Active cerebral/meningeal disease related to the underlying malignancy. Previous exposure to CD228-targeted therapy, vedotin or an MMAE-containing agent, or any taxane containing regimen for advanced disease.

Melanoma subtypes including uveal, and mucosal are excluded. Chemotherapy, definitive radiotherapy, biologics, and/or other antitumor treatment with immunotherapy that is not completed 4 weeks prior to first dose of study intervention, or within 2 weeks prior to first dose of study intervention if the underlying disease has progressed on treatment

• Grade 3 or higher pulmonary disease unrelated to underlying malignancy. Previous history of non-infectious interstitial lung disease (ILD) or pneumonitis that required steroids, current ILD or pneumonitis, or suspected ILD or pneumonitis that cannot be ruled out by imaging at screening.

Other protocol specific criteria might apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | through 30 days after the last study treatment; approximately 6 months
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Number of participants with laboratory abnormalities | through 30days after the last study treatment; approximately 6 months
Number of participants with dose limiting toxicities | up to 28 days

SECONDARY OUTCOMES:
number of participants with antidrug antibodies | through 30 days after the last study treatment; approximately 6 months
  To be summarized using descriptive statistics
Pharmacokinetic (PK) parameter - Area under the curve (AUC) | Through 30 days after the last study treatment; approximately 6 months
  To be summarized using descriptive statistics
PK parameter - Maximum Concentration (Cmax) | Through 30 days after the last study treatment; approximately 6 months
  To be summarized using descriptive statistics
PK parameter - Time to maximum concentration (Tmax) | Through 30 days after the last study treatment; approximately 6 months
  To be summarized using descriptive statistics
PK parameter - Apparent terminal half-life (t1/2) | Through 30 days after the last study treatment; approximately 6 months
  To be summarized using descriptive statistics
PK parameter - Trough concentration (Ctrough) | Through 30 days after the last study treatment; approximately 6 months
  To be summarized using descriptive statistics
Objective response rate (ORR) | Up to approximately 1 year
  The proportion of participants with a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as assessed by the investigato
Duration of response (DOR) | Up to approximately 1 year
  The time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of progressive disease (PD) (based on radiographic assessments per RECIST v1.1) or death due to any cause
Progression-free survival (PFS) | Up to approximately 1 year
  The time from the start of study treatment to the first documentation of PD (per RECIST v1.1 as assessed by the investigator) or death due to any cause
Overall survival (OS) | Approximately 2 years
  The time from the start of study treatment to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (6):
  - The Angeles Clinic and Research Institue, A Cedars-Sinai Affiliate, Los Angeles, California
  - The Angeles Clinic And Research Institute, A Cedars-Sinai Affiliate, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - UCSF Medical Center, Investigational Pharmacy, San Francisco, California
  - The Angeles Clinic and Research Institue, A Cedars-Sinai Affiliate (Emergency Back-up only), Santa Monica, California
  - Sarah Cannon Research Institute at HealthONE - SCRI - PPDS, Denver, Colorado
- Gustave Roussy, Villejuif, Val-de-marne, France
- Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona], Spain
- Karolinska Universitetssjukhuset Solna, Solna, Stockholms LÄN [se-01], Sweden
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Sarah Cannon Research Institute UK, London, London, CITY of
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5901001